CLINICAL TRIAL: NCT03068663
Title: Characterization of Microbiota (intestinal, from Lungs, and Upper Airways) in Patients with Non-small Cell Lung Carcinoma: Exploratory Study
Brief Title: Microbiota and the Lung Cancer
Acronym: MICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Université d'Auvergne (Other); GREENTECH SA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-A01640-51
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; intestinal microbiota; lung microbiota; surgery; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 groups of patients will be follow :
  * Pchir : Non small cell lung carcinoma patients with an indication of immediate surgery.
  * Pct-chir : Non small cell lung carcinoma patients with an indication of neoadjuvant chemotherapy before the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pchir (Experimental): Non small cell lung carcinoma patients designated for immediate surgery. Intervention in this group is "sampling". The sampling will be done for:
  * blood and saliva: at consultations after inclusion in the study
  * faeces: day before the surgery
  * lung/tumour tissue, bronchoalveolar lavage: during surgery after lobectomy
  Interventions: Other: Sampling
- Pct-chir (Experimental): Non small cell lung carcinoma patients who will receive neoadjuvant chemotherapy before the surgery. Intervention in this group is "sampling". The sampling will be done for:
  * blood and saliva: 1st time at consultations after inclusion in the study, 2nd time at consultations after chemotherapy and before surgery
  * faeces: 1st time the day before the chemotherapy, 2nd time the day before the surgery
  * lung/tumour tissue, bronchoalveolar lavage: during surgery after lobectomy
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Patients will receive their standard treatments, surgery with/without chemotherapy. A patient intervention consists in taking samples of blood, saliva, faeces, lung/tumour tissue, and bronchoalveolar lavage fluid.

SUMMARY:
The subject is to study the lung microbiota and the one of upper airways (UAs) (much less studied than the intestinal microbiota) in 40 patients having lung cancer. 20 patients undergo only surgical treatment, while other half receives also chemotherapy. The idea is to explore changes in microbiota of the lung, upper UAs and intestine, and potentially find associations between them. These results will serve us as a base for the future study, focused on manipulation of the microbiota by prebiotics, probiotics or symbiotics and its effect on anti-cancer treatment tolerance and effectiveness.

DETAILED DESCRIPTION:
Lung cancer patients will be divided in two groups, a first one with patients undergoing both chemotherapy and surgery (Pct-chir), and the second one with patients only undergoing surgery (Pchir). Following inclusion, they will be given a 7-days alimentary survey, along with blood and saliva sampling (after buccodental examination and dental panoramic). The Pct-chir group will repeat the same procedure after the chemotherapy and before the surgery.

Day before the surgery, patients are asked to bring their faecal samples (in special box provided in advance) and the filled survey. During the operation the piece of lung tissue as well as the tumour (if the size enables it) will be sampled for further analysis. Lavage will be performed on the lung immediately after its resection.

Saliva, faecal sample, lung and tumour tissue, and lavage will be used for bacterial DNA extraction, followed by qPCR and sequencing analysis.

Lavage and blood samples will be analysed by flow cytometry and ELISA, to establish the immunological profile (interleukines, cell surface markers).

ELIGIBILITY:
Inclusion Criteria:

* non small cell lung carcinoma patient suitable for surgery, or chemotherapy followed by surgery
* BMI <29.9 kg/m²
* not taking antibiotics, corticosteroids and/or immunosuppressants at least during two months before inclusion
* not taking prebiotics, probiotics or symbiotics at least during two months before inclusion
* signing the written consent before enrollment in the study
* affiliation to the national health insurance (or system alike) according to the law from 9th August 2004

Exclusion Criteria:

* cognitive difficulties
* refusal of participation or inability to give a clear consent
* digestive or pulmonary infection of a long duration during the two months preceding the study (with antibiotic treatment)
* inflammatory digestive pathology
* concurrent treatment with experimental medication, participation in another clinical therapeutic study within 30 days
* presence of colostomy, total or partial gastrectomy
* previous esophageal surgery
* previous ORL (otho-rhino-laryngo) cancer treated by radiotherapy or surgery
* patient enable to follow the requirements of the study
* patient deprived of his rights by administrative or judicial decision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Difference in diversity of the lungs and upper airways microbiota | 1.5 - 4.5 months
  The analysis of the diversity will be performed by DNA sequencing and qPCR on the different samples (saliva, bronchoalveolar lavage and lung tissue fragments).

SECONDARY OUTCOMES:
Effect of chemotherapy on microbiota (by comparing before and after chemotherapy) | 3.5-4.5 months
  Difference in the proportion of the Firmicutes phylum between UAs and lungs, and difference in the proportion of most abundant bacterial phyla between three types of samples (saliva, lung tissue, faecal samples), all analysed by qPCR and sequencing.
inflammatory status | 1.5 - 4.5 months
  dosage of plasmatic cytokines and interleukins (ELISA or luminex)
effect of microbiota on pulmunary immune cells | 1.5 - 4.5 months
  characterization of immune cells on lung/tumor sample and bronchoalveolar lavage fluid (flow cytometry and/or immunohistochemistry)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Paule Vasson, Pr, Study Director — Equipe ECREIN, CLARA, CRNH Auvergne; INRA, UMR 1019.; Edith Filaire, Pr, Study Director — CIAMS, Université Paris-Sud, Université Paris-Saclay, Université Orléans; Annick Bernalier-Donadille, Dr, Study Director — Equipe MINHOS, UR 454 Microbiologie, INRA; Rea Bingula, Ph.D., Study Director — Equipe ECREIN, CLARA, CRNH Auvergne; INRA, UMR 1019; Marc Filaire, MD, Pr, Principal Investigator — Service de Chirurgie Thoracique, Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, puy de dôme, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montassier E, Gastinne T, Vangay P, Al-Ghalith GA, Bruley des Varannes S, Massart S, Moreau P, Potel G, de La Cochetiere MF, Batard E, Knights D. Chemotherapy-driven dysbiosis in the intestinal microbiome. Aliment Pharmacol Ther. 2015 Sep;42(5):515-28. doi: 10.1111/apt.13302. Epub 2015 Jul 6. PMID 26147207
- [Derived] Bingula R, Filaire E, Molnar I, Delmas E, Berthon JY, Vasson MP, Bernalier-Donadille A, Filaire M. Characterisation of microbiota in saliva, bronchoalveolar lavage fluid, non-malignant, peritumoural and tumour tissue in non-small cell lung cancer patients: a cross-sectional clinical trial. Respir Res. 2020 May 25;21(1):129. doi: 10.1186/s12931-020-01392-2. PMID 32450847